CLINICAL TRIAL: NCT00371800
Title: The Effect of Cinnamon on HbA1c Among Adolescents With Type I Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17648
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Cinnamon; Type 1 Diabetes; Adolescent; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: cinnamon

SUMMARY:
the purpose of this study is to determine if cinnamon improves glucose control among adolescents with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Widespread achievement of glucose control remains an elusive goal for adolescents with Type 1 diabetes. Previous research has suggested that cinnamon may be effective at improving glucose control in type 2 diabetes. To date, no research has investigated the effect of cinnamon on type 1 diabetics. If the addition of a simple, natural, pill to a standard insulin regimen can significantly improve glucose control, the clinical implications would be substantial.

Comparison: Using a prospective, double-blind, placebo-controlled design, 72 adolescent type I diabetics were treated with cinnamon (1 gram/day) or an equivalent appearing placebo for 90 days. HbA1c, total daily insulin intake, and adverse events were recorded and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 1 diabetes for > 18 months prior to enrollment,
2. Age 13-18 years at the time of enrollment
3. Presenting to the clinic for routine care,
4. No hospital admissions for medical or psychiatric reasons in the 12 months prior to enrollment,
5. Accessible by phone,
6. Not pregnant.

Exclusion Criteria:

(1) Pregnant

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72
Dates: Start 2005-10; Study Completion 2006-05

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
Total Daily Insulin
Carbohydrate/insulin dose
Hypoglycemic events
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Casella, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States